CLINICAL TRIAL: NCT04878250
Title: A Phase II Study Investigating Preoperative Bintrafusp Alfa in Operable Urothelial Carcinoma of the Bladder
Brief Title: Preoperative Bintrafusp Alfa in Operable Urothelial Carcinoma of the Bladder
Acronym: PEBBLE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEBBLE
Record Dates: First submitted 2021-04-30; First posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Transitional Cell Carcinoma; Bladder Cancer
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — bintrafusp alfa protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bintrafusp alfa (Experimental)
  Interventions: Drug: Bintrafusp alfa

INTERVENTIONS:
Drug: Bintrafusp alfa — 4 doses of bintrafusp alfa (1200mg flat dose) administered intravenously at 14 day intervals before undergoing radical cystectomy.

SUMMARY:
PEBBLE is an open-label, international, multicentre, window of opportunity phase II trial that aims to evaluate the effects of short-term preoperative therapy with bintrafusp alfa in patients with histologically confirmed urothelial carcinoma requiring radical surgery with bilateral pelvic lymph node dissection. Eligible patients will receive 4 doses of bintrafusp alfa (1200mg flat dose) at 14 day intervals before undergoing radical surgery. Patients will attend study visits at 6, 12 and 24 weeks following their surgery. After the 24-week post-surgical visit, patients will enter a follow up phase during which they will be contacted annually for 2 years after their surgery to collect survival and disease status data. The efficacy of bintrafusp alfa will be assessed on CT/MRI scan images and tumour tissue samples collected at baseline and after treatment with bintrafusp alfa.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Ability to comply with the protocol
3. Age ≥ 18 years
4. Histopathologically confirmed urothelial carcinoma (T2-T4aN0-1M0) of the bladder where radical cystectomy with bilateral pelvic lymph node dissection is indicated. Patients with "variant histology" such as micropapillary, plasmocytoid, nested, sarcomatoid, microcystic, squamous and adeno variants of urothelial carcinoma are required to have more than 50% of tumor tissue with transitional cell pattern.
5. Residual disease after TURBT or endoscopy (surgical opinion, cystoscopy or radiological presence).
6. Fit and planned for surgery (according to local guidelines).
7. N0-1 and M0 disease CT or MRI (within 4 weeks of enrolment). Patients with N2 disease on cross sectional imaging are excluded from the study.
8. Representative formalin-fixed paraffin embedded (FFPE) tumour samples with an associated pathology report that are determined to be available and sufficient for central testing.
9. Patients who refuse neoadjuvant cisplatin-based chemotherapy or in whom neoadjuvant cisplatin-based therapy is not appropriate.
10. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
11. Negative serum pregnancy test within 14 days of Day 1 Cycle 1 for female patients of childbearing potential.
12. Highly effective method of contraception throughout the study until 2 months after the last dose of bintrafusp alfa for female patients of childbearing potential and 4 months after the last dose of bintrafusp alfa for male patients.
13. Adequate haematologic and end-organ function within 4 weeks prior to the first study treatment.

Exclusion Criteria:

1. Pregnant and lactating female patients.
2. Major surgical procedure within 4 weeks prior to enrolment or anticipation of need for a major surgical procedure during the course of the study other than for diagnosis.
3. Previous intravenous chemotherapy or immune therapy for bladder cancer.
4. Patients with prior allogeneic stem cell or solid organ transplantation.
5. Prior treatment with CD137 agonists, anti-CTLA-4, anti-programmed death-1 (PD-1), or anti-PD-L1 therapeutic antibody or pathway-targeting agents.
6. Has received any prior radiotherapy to the bladder.
7. Patients must not have had oral or intravenous (IV) steroids for 14 days prior to Cycle 1 Day 1. The use of inhaled corticosteroids, physiologic replacement doses of glucocorticoids (i.e., for adrenal insufficiency), and mineralocorticoids (e.g., fludrocortisone) is allowed at physiologic doses ≤ 10 mg/day of prednisone or equivalent.
8. Received therapeutic IV antibiotics within 14 days prior to enrolment (Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible).
9. Administration of a live, attenuated vaccine within 4 weeks prior to enrolment or anticipation that such a live, attenuated vaccine will be required during the study. Seasonal flu vaccines that do not contain a live virus are permitted.
10. Treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin [IL]-2) within 4 weeks or five half-lives of the drug, whichever is shorter, prior to enrolment.
11. Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 4 weeks prior to enrolment.
12. Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results, including significant liver disease (such as cirrhosis, uncontrolled major seizure disorder, or superior vena cava syndrome).
13. Malignancies other than urothelial carcinoma of the bladder within 3 years prior to enrolment with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, or ductal carcinoma in situ treated surgically with curative intent) or localized prostate cancer treated with curative intent and absence of prostate-specific antigen (PSA) relapse or incidental prostate cancer (Gleason score ≤ 3 + 4 and PSA < 10 ng/mL undergoing active surveillance and treatment naive).
14. Severe infections within 4 weeks prior to enrolment including but not limited to hospitalisation for complications of infection, bacteraemia, or severe pneumonia.
15. Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within 6 months prior to enrolment, unstable arrhythmias, or unstable angina.
16. History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organising pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan (History of radiation pneumonitis in the radiation field (fibrosis) is permitted).
17. Patients with uncontrolled Type 1 diabetes mellitus. Patients with Type 1 diabetes controlled on a stable insulin regimen are eligible.
18. Patients with active hepatitis infection (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C. Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
19. Positive test for HIV.
20. Patients with active tuberculosis.
21. History of autoimmune disease including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible. Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed. Patients with a history of autoimmune-related hypothyroidism, unless on a stable dose of thyroid-replacement hormone.
22. History of bleeding diathesis or recent major bleeding events (i.e. Grade ≥ 2 bleeding events in the 30 days prior to treatment
23. Has a diagnosis of immunodeficiency.
24. Receiving chronic systemic steroid therapy (in doses exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCRR) | Post - treatment with 4 cycles of bintrafusp alfa (1 cycle = 14 days)
  No microscopic evidence (pT0/Tis/Cis) of residual disease in the bladder based on histological evaluation of the resected bladder specimen collected during radical surgery

SECONDARY OUTCOMES:
Dynamic changes in TGFb, T-effector signatures and CD8 count measured in tumour samples. | Pre - and post - treatment with 4 cycles of bintrafusp alfa (1 cycle = 14 days)
Incidence, nature and severity of adverse events (AE) graded according to NCI-CTCAE v5.0 | From time of consent until the safety visit, an average of 22 weeks.
Disease free survival (DFS) defined as time between the date of enrolment to first evidence of relapse based on local investigator assessments or death, whichever occurs first. | Up to 2 years
Overall survival (OS) defined as the time between the date of enrolment and death due to any cause. | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Powles, Principal Investigator — Queen Mary University of London

IPD SHARING:
Plan to Share IPD: No